CLINICAL TRIAL: NCT06662474
Title: Evaluation of Cognitive Dysfunction in Patients with Breast Cancer Undergoing Systemic Therapy
Brief Title: Cognitive Impairment in Treated Breast Cancer Survivors: Possible Approaches
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Diana Ioana Boboc, Medical Oncologist, PhD Student, Investigator in Clinical Trials, Grigore T. Popa University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 445/28.05.2024
Record Dates: First submitted 2024-10-23; First posted 2024-10-29 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Cognitive Impairment; Chemobrain
Keywords: breast cancer; cognitive impairment; quality of life; intervention
MeSH Terms: conditions — Cognitive Dysfunction; Chemotherapy-Related Cognitive Impairment; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The present study is a prospective, multi-arm study at determining the cognitive impairment decline rate after 12 weeks of different interventions for each study group .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- cognitive stimulation arm (Active Comparator): will engage in exercises like sudoku, word games, and painting by numbers for 30 minutes per day, three days per week, for a duration of 12 weeks
  Interventions: Other: 1. cognitive stimulation
- psychoeducation and cognitive stimulation arm (Active Comparator): will engage in exercises like sudoku, word games, and painting by numbers for 30 minutes per day, three days per week, for a duration of 12 weeks and also hold open group meetings for psychoeducation (1 meeting every 2 weeks, 6 meetings in total).
  Interventions: Other: 2. psychoeducation and cognitive stimulation
- placebo (Placebo Comparator): is considered a control group, consisting of people who maintained their lifestyle up until their inclusion in the study without following additional measures
  Interventions: Other: 3. no intervention

INTERVENTIONS:
Other: 1. cognitive stimulation — sudoku, word games, and painting by numbers for 30 minutes per day, three days per week, for a duration of 12 weeks
  Arms: cognitive stimulation arm
Other: 2. psychoeducation and cognitive stimulation — sudoku, word games, and painting by numbers for 30 minutes per day, three days per week, for a duration of 12 weeks and also hold open group meetings for psychoeducation (1 meeting every 2 weeks, 6 meetings in total)
  Arms: psychoeducation and cognitive stimulation arm
Other: 3. no intervention — maintaines their lifestyle up until their inclusion in the study without following additional measures
  Arms: placebo

SUMMARY:
The investigators aim is to conduct a prospective study with three arms, involving non-metastatic breast cancer patients who underwent chemotherapy as part of their treatment and were on a form of hormone therapy at the time of study inclusion. The trial consists of identifying the presence of cognitive decline and following up on methods of preventing its accentuation. The goal of this clinical trial is to assess if psychoeducation and cognitive stimulation work to decrease the intensity of cognitive impairment. It aims to answer the following main questions:

* The implementation of such interventions improves both the dysfunction quantified by objective tests but also the individual's perception of it.
* The implementation changes the patients' quality of life. Researchers will compare three study groups, each with instructions to complete one of the related 12-week programs, to see if there are any changes.

Depending on the group in which the patient was randomly assigned, the interventions are :

* First group - will engage in exercises like sudoku, word games, and painting by numbers for 30 minutes per day, three days per week, for a duration of 12 weeks
* the second group will engage in exercises like sudoku, word games, and painting by numbers for 30 minutes per day, three days per week, for a duration of 12 weeks and also hold open group meetings for psychoeducation (1 meeting every 2 weeks, 6 meetings in total).
* Group 3 is considered a control group, consisting of people who maintained their lifestyle up until their inclusion in the study without following additional measures

DETAILED DESCRIPTION:
The trial consists of identifying the presence of cognitive decline and following up on methods of preventing its accentuation through psychoeducation and cognitive stimulation. The trial includes longitudinal assessments of some subjective perception markers and objective assessments of cognitive decline. Furthermore, the study will delve into the dynamics of these markers, revealing alterations in the psycho-affective state. The study aims to assess the impact of interventions on the cognitive decline associated with cancer and its treatment, as well as the role they can play in improving breast cancer patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* female patients aged 18 years or older
* histologically confirmed treated invasive non-metastatic HR positive
* provided written informed consent
* (ECOG) performance status 0 -2
* adequate hematologic functions
* the patients must have completed the treatment (surgery or chemotherapy) for a minimum of 6 months and a maximum of 3 years before enrolling in the study
* patients who received chemotherapy for at least 3 months, including both dose-dense regimens and those administered every 3 weeks, as part of their disease treatment.
* patients are considered eligible for study continuation if, in 1 month of screening procedures, the tests to identify depression and severe anxiety do not indicate a severe status for them.

Exclusion Criteria:

* history of neoplasia other than breast cancer
* brain metastases
* acute neurological diseases, neuro-degenerative or major psychiatric conditions such as stroke, autism, ADHD, Alzheimer's disease, Parkinson's disease, dementia, obsessive-compulsive disorder, post-traumatic stress disorder, schizophrenia, and those with a history of craniocerebral trauma
* associated pathologies who may receive any form of treatment
* the administration of psychotropic or pain medications in the II and III categories
* (ECOG) ≧3
* laboratory tests that contraindicate the administration of active oncological treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
presence of cognitive decline in breast cancer patients receiving systemic treatments | before initiating interventions
  using objective tests
rate of cognitive decline delay among those who implement prophylactic measures | from the moment the intervention was initiated until 6 months after the intervention
  using objective tests

SECONDARY OUTCOMES:
quality of life | from the moment the intervention was initiated until 6 months after the intervention
  The EORTC quality of life questionnaire (QLQ) is used for assessing the quality of life of cancer patients. A higher score indicates higher quality of life, while a lower a decrease of it.
psycho-emotional status - state of coping assessment | from the moment the intervention was initiated until 6 months after the intervention
  The investigators will be able to characterize the psycho-emotional status of the patients based on the scores obtained from evaluations using the Mental Adjustment Scale in Cancer. The scale (29 items) describes the state of coping that the patient has toward the disease The score is associated with the strength of behavior towards coping with cancer.
psycho-emotional status - assessment of disturbance | from the moment the intervention was initiated until 6 months after the intervention
  The investigators will be characterize the psycho-emotional status using DASS-21 R scales. The DASS-21 evaluates the negative emotion that a patient recognizes, represented by stress, anxiety, and depression.
  The severity of the affected psycho-emotional status increases the DASS-21 R scale score proportionally. The test associates the minimum score with a normal psychological response and categorizes an increase in scores based on the intensity of the symptoms.

IPD SHARING:
Plan to Share IPD: Undecided